CLINICAL TRIAL: NCT03246035
Title: A Prospective Randomized Pilot Trial to Reduce Readmission for Frail Elderly Patients With Acute Decompensated Heart Failure
Brief Title: Reducing Readmission for Frail Elderly Patients With Decompensated Heart Failure
Acronym: HFF-ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Collaborators: Canadian Association of Emergency Physicians (Industry)
Responsible Party: Principal Investigator, Jonathan Afilalo, Researcher, Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ADHF-ED-JGH
Record Dates: First submitted 2017-06-28; First posted 2017-08-11 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Heart Failure; Acute Decompensated Heart Failure; Fragility; Emergencies
Keywords: Acute Decompensated Heart Failure; Heart Failure; Frailty; Geriatrics; Self-care; Emergency Medicine; Cardiology; Patient Oriented Research
MeSH Terms: conditions — Heart Failure; Emergencies; Frailty | interventions — Control Groups; Standard of Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Standard Care) (Active Comparator): The control group will receive outpatient follow-up, medication advice and lifestyle guidance as prescribed at discharge from the ED or hospital.
  Interventions: Other: Control Group (Standard Care)
- Intervention Group (Experimental): The intervention will consist of contacting the patient 5 days post-discharge and arranging definitive outpatient follow-up and providing targeted medical and lifestyle advice based on deficient domains identified at baseline.
  Interventions: Behavioral: Intervention Group

INTERVENTIONS:
Behavioral: Intervention Group — For the intervention arm, a specialized heart failure nurse practitioner will contact the patient or their primary caregiver by telephone within 5 days post-discharge and send them an education packet by mail. During the telephone call, the nurse will (1) confirm the patient's scheduled follow-up appointment in cardiology, (2) provide recommendations for heart failure self-care behaviors that were found to be deficient at baseline. Patients will then be referred to a Geriatrics Assessment Team, who will provide individualized recommendations for frailty domains that were found to be deficient at baseline. The technique used to provide educational recommendations will be motivational interviewing.
  Arms: Intervention Group
Other: Control Group (Standard Care) — For patients randomized to the Control Group (Standard Care), they will receive their follow-up visits, medications, diet and physical activity advice as they normally would. This is the care they would receive even if they were not enrolled in the study
  Arms: Control Group (Standard Care)

SUMMARY:
A randomized study designed to determine whether telephone based interventions can prevent return hospital visits for elderly and frail patients with acute symptoms of heart failure. Specifically, the intervention will improve patients ability to monitor and address self care of heart failure at home.

DETAILED DESCRIPTION:
Acute decompensated heart failure (ADHF) is a common illness in Canadian emergency departments (ED). The frail subset of elderly patients with ADHF is challenging to treat, use a large proportion of available resources, and are at higher risk for complications, including readmission to hospital after discharge. The investigators believe that by improving access to follow-up, optimizing self-care, and addressing the various cognitive and physical limitations of frailty, it will be possible to improve quality of life and reduce readmission rates for frail patients with ADHF.

ELIGIBILITY:
Inclusion Criteria:

* Patients who presented to the ED and who are being discharged with a primary or secondary diagnosis of ADHF
* Age ≥ 65
* Frailty, defined as a FRAIL score >=3/5 or Clinical Frailty Scale (CFS) score >=5/9
* Informed consent provided by the patient or proxy

Exclusion Criteria:

* Significant dementia or active delirium
* Severe frailty, defined as a CFS score >=8/9
* Prohibitive language barrier
* Primary address outside of Quebec
* Patient deemed to be palliative or moribund by treating team

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
All-cause death, hospital readmission, or ED revisit | 90 days

SECONDARY OUTCOMES:
Rate of return visits to any ER for any medical issue | 30 days
  Number of times enrolled patient visits an emergency department for any medical issue, over the 90 day follow-up period.
Rate of admission to hospital at 90 days | 90 days
  Number of times the patient needs to be admitted to hospital for any medical issue, over the 3 month follow-up period.
Incidence of adverse effects from medication | 90 days
  Number of patients who experience unexpected side effects from their heart failure medications
Self-Care Index | 90 days
  Change in the Self-Care Heart Failure Index from enrollment to follow-up
Heart Failure Symptom Scale | 90 days
  Change in the 12 point Heart Failure Symptom Scale from enrollment to follow-up
Frailty Index | 90 days
  Change in the Frailty Index from enrollment to follow-up
Recruitment rate | 90 days
  The number of eligible of patients recruited into the study over a 3 month trial period
Attrition rate | 90 days
  The number of patients enrolled the study who choose to leave the study before completing the follow-up
Informed consent validation (qualitative) | 90 days
  Qualitative feedback from participants regarding the informed consent process
All-cause death, hospital readmission, or ED revisit | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Afilalo, FRCPC, Principal Investigator — Associate Professor
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Study Protocol: CODIM-MBM-17-052 — http://www.ladydavis.ca/en/jonathanafilalo — Pilot study protocol
- Available data/document: Informed Consent Form: CODIM-MBM-17-052 — http://www.ladydavis.ca/en/jonathanafilalo — Patient consent Caregiver consent French and English available